CLINICAL TRIAL: NCT02295917
Title: The Investigators Aim to Evaluate the Width of the Endometrial Myometrial Zone in Participants During Natural Menstrual Cycle by Using Specific Computerized Application on 3 Dimensions Sonographic Images of Their Uteri
Brief Title: Computerized Evaluation of the Endometrial Myometrial Junction During a Natural Menstrual Cyle.
Acronym: EMJ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Ronnie Tepper, Professor, Meir Medical Center
Other Study IDs: 0074-13-MMC
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Transvaginal sonography — Transvaginal sonography

SUMMARY:
The investigators aim to evaluate the width of the endometrial myometrial zone in participants during natural menstrual cycle by using specific computerized application on 3 dimensions sonographic images of their uteri.

DETAILED DESCRIPTION:
The uterine endometrium and the uterine myometrium have different acoustic characterization in transvaginal ultrasound(TVS).TVS can also demonstrate the interface between these tissues - the endometrial myometrial zone(EMJ) .This is optimally achieved in 3 dimensions images in a coronal section of the uterus.A specific computerized algorithm was developed in our unit by using MATLAB software for the quantitative measurements of the EMJ width in different uterine planes.The investigators aim to evaluate changes in the width of the EMJ in different uterine planes in participants during natural menstrual cycle .

ELIGIBILITY:
Inclusion Criteria:patients with regular menstrual cycles -

Exclusion Criteria:patients on contraceptive pills.patients after uterine surgery

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients referred for transvaginal sonography
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Changes in the width of the EMJ during natural cycle | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rami Aviram, MD, Principal Investigator — Meir Medical Center